CLINICAL TRIAL: NCT04705298
Title: Leveraging the Gut Microbiota in Pediatric Refractory Epilepsy: Safety and Feasibility of Oligofructose-enriched Inulin Supplementation for Dysbiosis and Seizure Control
Brief Title: Role of the Gut Microbiota in Pediatric Epilepsy
Acronym: EPBiome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, Maksim Parfyonov, Resident, Division of Neurology, British Columbia Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H19-01935
Record Dates: First submitted 2021-01-05; First posted 2021-01-12 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Drug Resistant Epilepsy
Keywords: Ketogenic Diet; Gut Microbiome; Inulin
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin 4 grams daily for ≤ age 6; or 8 grams daily for >6 years
  Interventions: Dietary Supplement: Placebo
- Prebiotic (Experimental): Oligofructose-enriched inulin 4 grams daily for ≤ age 6; or 8 grams daily for >6 years
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Oligofructose-enriched inulin. 4 grams daily for ≤ age 6; or 8 grams daily for >6 years
  Arms: Prebiotic
Dietary Supplement: Placebo — Maltodextrin 4 grams daily for ≤ age 6; or 8 grams daily for >6 years
  Arms: Placebo

SUMMARY:
Nearly a third of children with epilepsy are refractory to pharmacotherapy. The ketogenic diet (KD) is a highly effective alternative therapy reducing seizure frequency by 50% in more than half of treated children. The exact mechanisms of KD remain poorly understood, and recent studies have implicated the gut microbiota (GM). This pilot study aims to determine the feasibility of a 12-week dietary intervention with prebiotic fiber in children with epilepsy. The investigators hypothesize that consumption of inulin will alter gut microbiota and may have effects on seizure frequency.

ELIGIBILITY:
* Inclusion Criteria:

  * Children with epilepsy:

    1. Age 2-18.
    2. Attended the epilepsy clinic for a minimum of 6 months.
    3. On a stable number and type of medications for 4 weeks.
    4. Have not previously been on the ketogenic diet.
  * Healthy controls:

    1. Aged 2-18.
    2. Immunocompetent.
    3. No medical comorbidities (e.g. autoimmune, metabolic, cardiovascular, renal, or gastrointestinal conditions).
* Exclusion Criteria:

  1. Health conditions such as disorders of fatty acid transport and oxidation, porphyria, and pancreatitis, Glucose transporter 1 deficiency, pyruvate dehydrogenase deficiency, diabetes, and other autoimmune diseases.
  2. Presence of HIV infection, chronic wound infection, or osteomyelitis
  3. Presence of or treatment for periodontal infection
  4. Inflammatory bowel disease, chronic diarrhea, current Clostridium difficile infection
  5. Treatment with immunosuppressive agents in the past 6 months
  6. Significant changes in dietary intake (i.e. excluded sugar, lactose or gluten from their diet, started consuming a vegetarian or vegan diet) over the past 6 months.
  7. Gastrointestinal illness in the past month or food intolerances leading to gastrointestinal symptoms.
  8. Use of antibiotics in the 3 months preceding the study.
  9. Use of probiotic or prebiotic supplements in the month preceding the study.
  10. Consumption of probiotic yoghurt in the past 2 weeks.
  11. Use of laxatives, proton pump inhibitors, or gastric motility medications in the month preceding the study.
  12. History of allergic reaction or intolerance of maltodextrin or inulin.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in alpha and beta bacterial diversity measures in stool | 12 weeks
  Compare the effect of oral inulin vs. placebo on alpha and beta bacterial diversity in the stool of children undergoing ketogenic diet therapy for epilepsy
Change in Short Chain Fatty Acid (SCFA) levels in stool | 12 weeks
  Compare the effect of inulin vs. placebo on SCFA levels in the stool of children undergoing ketogenic diet therapy for epilepsy

SECONDARY OUTCOMES:
Seizure frequency | 12 weeks
  Trends in seizure frequency during inulin treatment compared to pre-treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia